CLINICAL TRIAL: NCT00715195
Title: Evaluation of Improving Quality of Life of Fibromyalgia Patients Treated With a Plurifocal Program : a Controlled Study With 12 Months Monitoring.
Brief Title: Improving Quality of Life of Fibromyalgia Patients
Acronym: Aquavip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P051029
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2013-11

CONDITIONS: Fibromyalgia
Keywords: Cognitive behavioral; Long-term study; Education
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cognitive-behavioral therapy : 50 patients planned
  Interventions: Behavioral: Plurifocal educational program
- 2 (No Intervention): 50 patients planned

INTERVENTIONS:
Behavioral: Plurifocal educational program — intensive group program of 8 weeks, including, in addition to the briefing, measures and exercises for the implementation of the principles of managing fibromyalgia, and cognitive-behavioral therapy
  Arms: 1

SUMMARY:
Comparison of two treatments of fibromyalgia; the QOL score should improve rather and, twelve months after the end of the program, remain higher in "Plurifocal educational group" than in control group

DETAILED DESCRIPTION:
Comparing two forms of non-drug treatment of fibromyalgia: "Information" (an information group session on the fibromyalgia management modalities) versus "Plurifocal educational program " (intensive group program of 8 weeks, including, in addition to the briefing, measures and exercises for the implementation of the principles of managing fibromyalgia, and cognitive-behavioral therapy).

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia Patients according to the criteria of the American College of Rheumatology defined by:

  * diffuse pain evolving for over three months
  * pain on palpation of at least 11 of the 18 sites listed
* age between 18 and 65
* FIQ Score higher than 35/100 at inclusion
* Ability to respond to questionnaires
* monitoring possibility for at least a year
* Affiliation to the French Health System (social security)

Exclusion Criteria:

* Association with chronic pain from other sources which can interfere with fibromyalgia assessment
* Inability to follow the full educational program
* previous participation in an educational program of same nature
* psychological disorder (personality disorder or behaviour, schizophrenia), preventing participation in the program group

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2007-09; Primary Completion 2011-12 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Score of the Fibromyalgia Impact Questionnaire, at one month and twelve months after program end | one month and twelve months after program end

SECONDARY OUTCOMES:
Pain Numeric scale,Number of tender points, Sleep quality numeric scale,Pain Impact Questionnaire ANAES,STAI-Y anxiety questionnaire,Beck Depression Index II,Coping Strategy Questionnaire,Multidimensional self-assessment(SF36, PSOCQ) | one , six and twelve months after program end

CONTACTS AND LOCATIONS:
Overall Officials: Guy COICHARD, MD Ph, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Saint Antoine, Paris, France